CLINICAL TRIAL: NCT02997410
Title: Effect of High-frequency Bio-oxidative Ozone Therapy for Masticatory Muscle Pain: a Double-blind Randomized Clinical Trial
Brief Title: Ozone Therapy for Masticatory Muscle Pain (OTMMP)
Acronym: OTMMP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Tamer Celakil, Research Assistant, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TCelakil
Record Dates: First submitted 2016-12-13; First posted 2016-12-20 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Orofacial Pain; Temporomandibular Joint Disorders
Keywords: Ozone
MeSH Terms: conditions — Facial Pain; Temporomandibular Joint Disorders | interventions — Dental Care; Occlusal Splints

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ozone (Experimental): Ozone application to the greatest points of pain in the related muscle, 3 times per week for 2 weeks
  Interventions: Device: Ozone
- Placebo (Placebo Comparator): Sham ozone application to the greatest points of pain in the related muscle, 3 times per week for 2 weeks
  Interventions: Device: Placebo (for Ozone)
- Occlusal splint (Experimental): Occlusal splint use every night over a period of 4 weeks.
  Interventions: Device: Dental treatment with occlusal splint

INTERVENTIONS:
Device: Ozone
  Other Names: OzonytroneX
  Arms: Ozone
Device: Placebo (for Ozone)
  Arms: Placebo
Device: Dental treatment with occlusal splint
  Arms: Occlusal splint

SUMMARY:
This study investigates the efficacy of bio-oxidative ozone application in the treatment of TMD of muscular origin.

DETAILED DESCRIPTION:
Ozone is a natural pale blue gas that can be found in the atmosphere. Medical grade ozone is a powerful oxidizing agent which can be produced commercially in ozone generators. Ozone can have effects on blood components and positively affect oxygen metabolism, cell energy, immunomodulation and microcirculation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of myofascial pain according to the Research Diagnostic Criteria for Temporomandibular Disorder (RDC/TMD)
* Natural posterior occlusion.

Exclusion Criteria:

* Any TMJ internal derangement
* Inflammatory connective tissue disease
* Psychiatric problem
* Tumour
* Hearth disease or pacemaker
* Pregnancy
* Other orofacial region disease symptoms (e.g. toothache, neuralgia, migraine)
* Treatment or medication use for headache or bruxism in the last 2 years
* Local skin infection over the masseter or temporal muscle

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-12; Primary Completion 2017-06 (Actual); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Pain Values (kg/cm2) on the Pressure pain threshold measurement (PPT) using a Pressure Algometry at 1 month | Change from Baseline Pain Values (kg/cm2) at 1 month
  Patient-reported pain intensity data when the feeling of pressure become painful, at which time the pressure is stopped. Measurements were separated by 30-s rest periods.
Change From Baseline in Pain Values (kg/cm2) on the Pressure pain threshold measurement (PPT) using a Pressure Algometry at 3 months | Change from Baseline Pain Values (kg/cm2) at 3 months
  Patient-reported pain intensity data when the feeling of pressure become painful, at which time the pressure is stopped. Measurements were separated by 30-s rest periods.
Change From Baseline in Pain Scores on the Visual Analog Scale at 1 month | Change from Baseline Pain Scores at 1 month
  The measurement of subjective pain intensity is done using a 100-mm visual analogue scale.
Change From Baseline in Pain Scores on the Visual Analog Scale at 3 months | Change from Baseline Pain Scores at 3 months
  The measurement of subjective pain intensity is done using a 100-mm visual analogue scale.

SECONDARY OUTCOMES:
Functional examination | Baseline, 1 month and 3 months
  Functional examination is based on Research Diagnostic Criteria for Temporomandibular Disorder (RDC/TMD) including extra-oral and cervical muscle pains, joint pains, mouth openings, lateral excursions and protrusion. Vertical and horizontal movements are measured with a plastic millimetre-scale ruler. Participants are asked to report any pain during muscle and joint palpation, and this information is recorded using a verbal scale: 0, no pain; 1, mild pain; 2, moderate pain; and 3, severe pain.

REFERENCES:
- [Background] Dogan M, Ozdemir Dogan D, Duger C, Ozdemir Kol I, Akpinar A, Mutaf B, Akar T. Effects of high-frequency bio-oxidative ozone therapy in temporomandibular disorder-related pain. Med Princ Pract. 2014;23(6):507-10. doi: 10.1159/000365355. Epub 2014 Sep 3. PMID 25196631
- [Background] Daif ET. Role of intra-articular ozone gas injection in the management of internal derangement of the temporomandibular joint. Oral Surg Oral Med Oral Pathol Oral Radiol. 2012 Jun;113(6):e10-4. doi: 10.1016/j.tripleo.2011.08.006. Epub 2012 Feb 28. PMID 22677023